CLINICAL TRIAL: NCT05168839
Title: Intraoperative Indocyanine Green Fluorescence Angiography in Colorectal Surgery to Prevent Anastomotic Leakage: a Single-blind Phase III Multicenter Randomized Controlled Trial (Intergroup FRENCH-GRECCAR Trial)
Brief Title: Intraoperative Indocyanine Green Fluorescence Angiography in Colorectal Surgery to Prevent Anastomotic Leakage
Acronym: FLUOCOL-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-582
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer
Keywords: Anastomotic leakage; Colorectal surgery; fluorescence angiography; Indocyanine green; Colic surgery; Complication; Prevention; Rectal surgery
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLUO+ (Experimental): Experimental arm = surgery with IOFA.
  In the experimental arm, cancer resection and anastomosis will be performed after assessment of descending colon perfusion using intravenous injection of indocyanine green 0.1ml/kg.
  Interventions: Drug: FLUO+ : Intraoperative fluorescence angiography (IOFA) with indocyanine green (ICG).
- FLUO- (No Intervention): Control arm = Surgery without IOFA.
  In the control arm, cancer resection and anastomosis will be performed without intraoperative fluorescence angiography.

INTERVENTIONS:
Drug: FLUO+ : Intraoperative fluorescence angiography (IOFA) with indocyanine green (ICG). — In the experimental arm (FLUO+), at least one 0.1mg/kg Infracyanine® bolus will be injected intravenously by the anesthesiologist.
  The detection of indocyanine green in the proximal colon segment will be done open or intracorporeally using a dedicated infrared camera.
  A surgical film describing the injection technique and fluorescence detection will be presented during the study set-up visits.
  An additional injection is allowed at the surgeon's discretion if necessary (change of anastomosis site). The time from injection to indocyanine green detection and any adverse events will be recorded.
  Arms: FLUO+

SUMMARY:
Colorectal cancer (CRC) is the fourth most commonly diagnosed cancer in the world and the third in France. Its incidence is steadily rising in developing nations. Anastomotic leak (AL) is a major problem in colorectal surgery affecting at least 7% of patients operated on for left colonic cancer. It is the most feared complication after colorectal anastomosis, associated with mortality, prolonged hospitalization, impaired health related quality of life (HRQoL) and increased health care costs. Intraoperative fluorescence angiography (IOFA) with indocyanine green (ICG) may help preventing AL. Available studies on the effects of IOFA with ICG are heterogeneous and randomized controlled trial are scarce. Our aim is to demonstrate that IOFA with ICG could lead to a reduction of AL rate after left-sided or low anterior resection with anastomosis for CRC.

The FLUOCOL-1 study is the first national, multicenter, single blind, randomized, 2-arm, phase III superiority clinical trial. The primary endpoint is the occurrence of an AL 90 days post-operation. AL is defined as any anastomotic dehiscence with leakage into the pelvic cavity diagnosed upon imaging or at surgical exploration or any isolated pelvic organ-space infection with no evidence of fistula as defined by the International Study Group of Rectal Cancer.

The study population will be made of adult patients with left-sided or high rectal cancer scheduled to undergo elective left colectomy or high rectal resection (by open, laparoscopy or robotic surgery) and with expected stapled or hand-sewn intraperitoneal anastomosis. The exclusion criteria are mainly an emergent surgery; rectal cancer requiring total mesorectal excision and anastomosis expected below the peritoneal reflection; CRC requiring total or subtotal colectomy; CRC requiring transverse colectomy; recurrent CRC and locally advanced colorectal cancer requiring multi-visceral excision.

A total of 1010 patients will be necessary (39 patients in each centre during 36 months). An interim analysis for efficacy and futility is scheduled when half of the participants will have been recruited.

In case of positive results favoring IOFA, this study would define the use of IOFA as a standard of care in colorectal surgery. At the patient level, a significantly lower rate of AL will reduce hospital stay and stoma rate, and will ensure improved postoperative recovery, faster return to normal activity and better long-term oncologic outcomes.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the fourth most commonly diagnosed cancer in the world and the third in France. Its incidence is steadily rising in developing nations. Anastomotic leak (AL) is a major problem in colorectal surgery affecting at least 7% of patients operated on for left colonic cancer. It is the most feared complication after colorectal anastomosis, associated with mortality, prolonged hospitalization, impaired health related quality of life (HRQoL) and increased health care costs. Intraoperative fluorescence angiography (IOFA) with indocyanine green (ICG) may help preventing AL. Available studies on the effects of IOFA with ICG are heterogeneous and randomized controlled trial are scarce. Our aim is to demonstrate that IOFA with ICG could lead to a reduction of AL rate after left-sided or low anterior resection with anastomosis for CRC.

The FLUOCOL-1 study is the first national, multicenter, single blind, randomized, 2-arm, phase III superiority clinical trial. The primary endpoint is the occurrence of an AL 90 days post-operation. AL is defined as any anastomotic dehiscence with leakage into the pelvic cavity diagnosed upon imaging or at surgical exploration or any isolated pelvic organ-space infection with no evidence of fistula as defined by the International Study Group of Rectal Cancer.

The study population will be made of adult patients with left-sided or high rectal cancer scheduled to undergo elective left colectomy or high rectal resection (by open, laparoscopy or robotic surgery) and with expected stapled or handsewn intraperitoneal anastomosis. The exclusion criteria are mainly an emergent surgery; rectal cancer requiring total mesorectal excision and anastomosis expected below the peritoneal reflection; CRC requiring total or subtotal colectomy; CRC requiring transverse colectomy; recurrent CRC and locally advanced colorectal cancer requiring multi-visceral excision.

The 26 participating centres are equipped with a scope with near-infrared (NIR) light source allowing real-time ICG perfusion assessment. The co-investigators are experienced digestive surgeons trained to work with and without IOFA. They have considerable experience in working together on research projects and have a proven track-record of efficacy. Moreover, this study will receive valuable support from the Surgery Research Network (FRENCH) and the Surgical Research on Rectal Cancer Group (GRECCAR), which have proved their ability to recruit patients into various multicentric studies and with which the FLUOCOL-1 project has been discussed.

The duration of participation for each patient is 90 days. The 3 study visits are superimposed to the schedule of standard of care (V1: pre-operation visit of selection and inclusion; Surgery; V2: 30-day post-operation visit and V3: 90-day post-operation visit).

The surgeon will do the 1:1 randomization between V1 and the day before surgery (D-30 to D-1). To reduce the risk of bias, patients will be blinded to the study group and the randomization will be stratified on participating centres, Body Mass Index (BMI), physical status classification score (=ASA score), preoperative treatment and tumor location. Patient will be assigned in the intervention (IOFA) or the control group (no IOFA).

At the exception of the information given on the study to the patient, the gathering of the written consent, the randomization and the HRQoL questionnaires, the patient will be treated following standard of care. Study data are the data systematically collected in the patient medical file except for the HRQoL questionnaires that will be collected under the supervision of a research technician financed by the study. The technician will capture the study data and the de-identified pdf version of the medical reports (consultations and hospitalizations) in the electronic Case Report Form (eCRF) after every visit.

A total of 1010 patients will be necessary (39 patients in each centre during 36 months). An interim analysis for efficacy and futility is scheduled when half of the participants will have been recruited.

The ICG will be graciously provided by the manufacturer (SERB). An investigator meeting will be organized twice a year during the annual GRECCAR and FRENCH meetings. Newsletters will be sent every 3 months.

In case of positive results favoring IOFA, this study would define the use of IOFA as a standard of care in colorectal surgery. At the patient level, a significantly lower rate of AL will reduce hospital stay and stoma rate, and will ensure improved postoperative recovery, faster return to normal activity and better long-term oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years)
* Scheduled to undergo elective left colectomy or high rectal resection for cancer with intraperitoneal anastomosis.
* Signed consent
* Affiliated to the French social security system (CMU included).

Exclusion Criteria:

* Emergent surgery.
* Rectal cancer requiring total mesorectal excision and anastomosis below the peritoneal reflexion.
* Colon cancer requiring total or subtotal colectomy defined as a right colectomy extended to the splenic flexure or more).
* Colon cancer requiring transverse colectomy.
* Recurrent colorectal cancer.
* Locally advanced colorectal cancer requiring multi-visceral excision.
* History of colectomy.
* Associated concomitant resection of other organ (liver, etc.).
* Previous pelvic radiotherapy for pathology unrelated to diagnosis with colon cancer e.g. treatment for prostate cancer.
* Inflammatory bowel disease.
* History of known allergy to indocyanine.
* Pregnant patients.
* Refusal to participate or inability to provide informed consent.
* Protected adults (individuals under guardianship by court order).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage 90 days after surgery | 90 days after surgery
  The primary outcome is the occurence of an anastomotic leakage during the 90 days following surgery.
  Anastomotic leakage is defined as any clinical signs of leakage diagnosed by radiological examination or surgical exploration, or as any isolated pelvic organ infection without leakage evidence, as defined by the International Rectal Cancer Study Group.

SECONDARY OUTCOMES:
Change in planned anastomotic site. | During surgery
  Change in planned anastomosis during surgery is defined as any decision change on perfusion assessment such as modifying the initially planned transection level of the descending colon or refashioning anastomosis including the decision to undertake a permanent stoma rather than an anastomosis.
Rate of patients with a defunctioning stoma. | Surgery time.
  The rate of defunctioning stoma created in the initial surgery as a temporary diverting pathway will be calculated.
Overall 30-day postoperative morbidity. | 30 days after surgery.
  Overall 30-day postoperative morbidity is defined and classified according to the Clavien-Dindo classification.
Overall 90-day postoperative morbidity. | 90 days after surgery.
  Overall 90-day postoperative morbidity is defined and classified according to the Clavien-Dindo classification.
Mortality rate. | 90 days after surgery.
  90-day postoperative mortality.
Hospital length of stay. | End of hospital stay.
  Postoperative length of hospital stay.
Postoperative reintervention. | 90 days after surgery.
  Postoperative reintervention number and type within 90 days.
Quality of life assessment. | 90 days after surgery.
  Health related quality of life is assessed using the quality of life questionnaires : QLQ-C30 and QLQ-CR29 at baseline and 90 days post-operation.
  The QLQ-C30 is a patient self-rating questionnaire (30 questions) that measures physical, role, social, emotional, and cognitive functions as well as overall QoL. Scores can be linearly transformed to provide a score from 0 to 100 REF. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
  The QLQ-CR29 (Quality of life of rectal cancer patients with 29 questions) has five functional and 18 symptom scales. It contains four subscales (urinary frequency (UF), blood and mucus in stool (BMS), stool frequency (SF), and body image (BI)) and 19 single items. The score can range from 0 to 100.
  Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Medico-economic analysis | 90 days after surgery.
  The medico-economic analysis takes into consideration health care costs up until 90 days post-operation.

CONTACTS AND LOCATIONS:
Locations (32):
- France (32):
  - Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - CH Annecy, Annecy
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Bourgoin-Jallieu, Bourgoin
  - University Hospital of Dijon, Dijon
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre lyonnais de chirurgie digestive, Lyon
  - Centre Hospitalier Lyon-Sud, Lyon
  - Hôpiatl Européen, Marseille
  - Hôpital La Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Nord AP-HM, Marseille
  - Hôpital St Joseph Marseille, Marseille
  - CHU de Nancy, Nancy
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Bicêtre, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier de Pontoise, Pontoise
  - Hôpital Robert Debré, Reims
  - Ch Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Santé Atlantique, Saint-Herblain
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Clinique TIVOLI, Toulouse
  - Centre Hospitalier de Tours, Tours
  - Institut cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wojcik M, Doussot A, Manfredelli S, Duclos C, Paquette B, Turco C, Heyd B, Lakkis Z. Intra-operative fluorescence angiography is reproducible and reduces the rate of anastomotic leak after colorectal resection for cancer: a prospective case-matched study. Colorectal Dis. 2020 Oct;22(10):1263-1270. doi: 10.1111/codi.15076. Epub 2020 May 18. PMID 32306516